CLINICAL TRIAL: NCT01312987
Title: Improving Nutrition and Health Outcomes in Intibuca, Honduras
Brief Title: Improving Nutrition and Health Outcomes in Intibuca, Honduras (MANI I)
Acronym: MANI I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shoulder to Shoulder (Other)
Collaborators: The Mathile Institute for the Advancement of Human Nutrition (Other)
Responsible Party: Jeff Heck, MD, Executive Director, Shoulder to Shoulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MANI I, Shoulder to Shoulder
Record Dates: First submitted 2011-03-05; First posted 2011-03-11 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Malnutrition; Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition intervention (Experimental): Receives a month's supply of the nutrition supplement, Plumpy'doz®, in addition to food voucher for each month. Participants were also allowed to attend monthly educational sessions.
  Interventions: Dietary Supplement: Lipid-based nutritional supplement
- Control (No Intervention): Receives food vouchers each month.
  Interventions: Dietary Supplement: Lipid-based nutritional supplement

INTERVENTIONS:
Dietary Supplement: Lipid-based nutritional supplement — After gradual introduction of the lipid-based nutritional supplement, daily dose per child is as follows:
  3 teaspoons 3 x day for children younger than 12 months 4.5 teaspoons 3 x day for children older than 12 months
  Other Names: Plumpy'doz®

SUMMARY:
The purpose of this research study is to assess what impact an integrated educational and feeding intervention delivered to infants and children has on growth (weight and height), development (cognitive and gross motor), nutrition (dietary behaviors, food insecurity, and micronutrient status - folate, iron, zinc, vitamin A, vitamin D), and morbidity (respiratory and diarrheal) outcomes. A randomized community trial was used to implement a nutrition intervention program consisting of monthly education sessions, a lipid-based nutrition supplement, and food vouchers for local staples.

ELIGIBILITY:
Inclusion Criteria:

* All healthy children between the ages of 5-18 months old and their mothers who are residents of the municipalities of Santa Lucia, Magdalena and San Antonio who do not present any of the medical conditions listed in the exclusion criteria.
* Mothers have understood and signed consent forms to enable their children to participate in the study. They were willing to have their child participate in one or more blood draws, bi-monthly sessions: 1) nutrition classes and food voucher and lipid-based nutritional supplement and 2) height/weight monitoring, dietary intake questionnaire, and health outcome information. As well as the additional data assessments necessary to be considered active participants in the study.

Exclusion Criteria:

* Children with congenital anomalies, mental retardation, severe physical handicap, under-nutrition caused by medical conditions that contribute to under-nutrition such as heart disease, kidney failure, face and throat problems that interfere with swallowing, medical problems interfering with the absorption of food, chronic diseases such as tuberculosis, etc.
* Children with a known allergy to peanuts and eggs will also be excluded from the study, 30% of children with known allergies to nuts also have an allergy to eggs.
* Plans to move or change their place of residence outside of the study region in the next 2 months would make them ineligible.
* Mothers who are younger than 16 years of age will be excluded from the study. Women younger than 16 might not understand the consent process and the importance of following the guidelines established in the research, therefore we chose not to include this group as "eligible" participants.
* Children who are <= -2 standard deviations below the norm for z score for weight for age. These children are severely malnourished and need to be carefully followed under the supervision of a qualified health care provider.

Ages: 5 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height at 12 months | Baseline to month 12
  Participating children were measured by trained staff every month during the 12 month intervention.
Change from baseline in hemoglobin status at 12 months | Baseline to month 12
  Hemoglobin status was measured from blood samples taken by finger pricks at baseline, month 6, and month 12 of the intervention.
Change from baseline in serum transferrin status at 12 months | Baseline to month 12
  Serum transferritin was measured from blood samples taken by finger pricks at baseline, month 6, and month 12 of the intervention.
Change from baseline in C-Reactive Protein levels at 12 months | Baseline to month 12
  C-Reactive Protein was measured from dried blood spots collected at baseline, month 6, and month 12 of the intervention.
Change from baseline in weight at 12 months | Baseline to month 12
  Participating children were weighed by trained staff every month during the 12 month intervention.

SECONDARY OUTCOMES:
Change from baseline in zinc levels at 12 months | Baseline to month 12
  Zinc status was measured from blood samples taken by finger pricks at baseline, month 6, and month 12 of the intervention.
Change from baseline in food insecurity status at 12 months | Baseline to month 12
  Assessment teams administered a scored questionnaire at baseline and month 12 of the intervention.
Change from baseline in dietary intake based on 24-Hour Food Recall at 12 months | Baseline to month 12
  Assessment teams administered a 24-Hour Food Recall every month of the intervention.
Change from baseline in various health outcomes at 12 months | Baseline to month 12
  Assessment teams administered a scored questionnaire every month of the intervention.
Change from baseline in acceptability of nutrition supplement at 12 months | Baseline to month 12
  Assessment teams administered a scored questionnaire at baseline, month 6, and month 12 of the intervention
Change from baseline in folate status at 12 months | Baseline to month 12
  Folate status was measured from blood samples taken by finger pricks at baseline, month 6, and month 12 of the intervention.
Change from baseline in vitamin B12 status at 12 months | Baseline to month 12
  Vitamin B12 was measured from blood samples taken by finger pricks at baseline, month 6, and month 12 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Heck, MD, Principal Investigator — Shoulder to Shoulder